CLINICAL TRIAL: NCT01472445
Title: Vitamin D and Breast Cancer: Does Weight Make a Difference?
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Melinda Telli (Other)
Responsible Party: Sponsor-Investigator, Melinda Telli, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-21034; SU-09262011-8486 (Other: Stanford University); BRSADJ0024 (Other: OnCore)
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: Vitamin D; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-obese (Body Mass Index ≤ 25) (Experimental): Non-obese participants receive Vitamin D at 400 or 10,000 IU/day
  Interventions: Drug: Vitamin D
- Obese (Body Mass Index > 25) (Experimental): Obese participants receive Vitamin D at 400 or 10,000 IU/day
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D
  Other Names: cholecalciferol

SUMMARY:
This is a research study of the effect of Vitamin D on breast cancer. We hope to learn whether Vitamin D can change characteristics of certain genes in a breast cancer tumor that affect its growth. We believe some of these characteristics may be influenced by body weight.

DETAILED DESCRIPTION:
Vitamin D3 (cholecalciferol, colecalciferol) is one of type of vitamin D which is made by the skin when exposed to sunlight; it is also found in some foods and can be taken as a dietary supplement. It is used to treat and prevent vitamin D deficiency and associated diseases, including rickets. Vitamin D3 may have a role obesity and cancer biology. In the body, Vitamin D3 is metabolized to the active form 1,25-dihydroxycholecalciferol (calcitriol, 1,25-(OH)2vitamin D3).

This protocol is a randomized, controlled, and blinded clinical trial in obese and non-obese breast cancer patients in whom the effects of vitamin D supplementation will be evaluated in the neoadjuvant setting. Changes in biomarker expression levels in blood will be assessed from baseline to post-treatment (post-surgery).

Per protocol (see title), the treatment groups are defined as those participants with body mass index (BMI) ≤ 25 ("non-obese") and > 25 ("obese"). Within each treatment group, dose of Vitamin D3 was stratified between 400 IU/day (control) and 10,000 IU/day (experimental). All analyses were typically conducted between BMI cohorts stratified by Vitamin D3 dose.

Protocol Primary Objective: "To determine whether dietary vitamin D can reverse the negative effects of obesity and insulin resistance as reflected by changes in breast cancer gene expression patterns in obese and non obese subjects diagnosed with breast cancer."

Protocol Secondary Objectives: "To determine whether dietary vitamin D can reverse the negative effects of obesity and insulin resistance as reflected by serum biomarkers of insulin resistance and adipokine secretion in obese and non obese subjects diagnosed with breast cancer."

The following markers will be part of this study.

* Insulin-like growth factor-binding protein 3 (IGFBP-3) is a Vitamin D target, and the most abundant of 6 different IGFBPs. The insulin-like growth factors 1 and 2 (IGF-1 and IGF-2) binds to IGFBP-3 with high affinity, which helps lengthen the half-life of circulating IGFs in all tissues. Through this binding action, IGFBP-3 exerts anti-proliferative effects by blocking the ability of IGFs to activate the IGF-1 receptor (IGF1R, which stimulates cell proliferation). IGFBP-3 levels were assessed on the basis of mRNA levels.
* p21 [also known as p21Cip1; p21Waf1, cyclin-dependent kinase inhibitor 1 (CDKI1) or cyclin-dependent kinase (CDK)-interacting protein 1 (CDKIP1)] is the primary mediator of p53-dependent cell cycle arrest in response to DNA damage, and is a proliferation; apoptosis; and invasion biomarker. p21 is primarily associated with inhibition of CDK2, but is capable of inhibiting all cyclin/CDK complexes. p21 3 levels were assessed on the basis of mRNA levels.
* Matrix metalloproteinase-11 (MMP-11), aka Stromelysin-3 (SL-3), is involved in the breakdown of extracellular matrix in the disease processes of metastasis and arthritis, as well as various normal physiological processes, such as embryonic development, reproduction, and tissue remodeling. MMP-11 levels were assessed on the basis of mRNA levels.
* Ki-67 ("Antigen Identified By Monoclonal Antibody Ki-67", Antigen Ki67) is the protein produced by the gene MKI67, and is a nuclear protein that is associated with cellular proliferation and ribosomal RNA transcription. Ki-67 is a recognized biomarker for mitotic rate and cellular, but is absent in resting (quiescent) cells (Stage G0). In breast cancer, Ki67 identifies a subset of patients with ER-positive breast cancer that is highly proliferative, and who derive greater benefit from adjuvant chemotherapy. MKI67 levels were assessed on the basis of mRNA levels.
* ESR1 is the gene encoding estrogen receptor alpha (ERα), also known as NR3A1 (nuclear receptor subfamily 3, group A, member 1), and is a nuclear receptor that is activated by the sex hormone estrogen. ERα plays a role in the physiological development and function of a variety of organ systems to varying degrees, including the reproductive, central nervous, skeletal, and cardiovascular systems. Genetic polymorphisms in ESR1 have been associated with breast cancer. ESR1 levels were assessed on the basis of mRNA levels.
* Leptin is a stimulator of adipose stromal cell estrogen synthesis and a breast cancer growth promoter. Serum levels of leptin correlate with body mass index (BMI, a measure of obesity) and breast cancer risk. Leptin receptors are expressed by breast cancer cells and leptin can promote (regulate) breast cancer cell proliferation. Leptin levels were measured by Western blot or immunohistochemical (IHC) methodology.
* Adiponectin inhibits breast cancer growth. Adiponectin receptors are expressed by breast cancer cells and adiponectin can inhibit (regulate) breast cancer cell proliferation by stimulating apoptosis in estrogen receptor (ER)+ Breast cancer cells and suppressing estrogen-stimulated cell growth. Adiponectin levels were measured by Western blot or immunohistochemical (IHC) methodology.
* Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR) is a standard determination of insulin resistance based on fasting insulin and glucose levels.
* cRP (C-reactive protein) is an inflammation marker produced by the liver. High levels of CRP in the blood are indicative of a wide variety of conditions, including cancer. cRP levels were measured by Western blot or immunohistochemical (IHC) methodology.

ELIGIBILITY:
Inclusion Criteria:

* Women who have undergone a core needle biopsy demonstrating an operable breast cancer whom have not yet had any further therapy.
* No prior therapy for breast cancer.
* Age 18 years or older.
* Any menopausal status
* Planned surgical resection of breast cancer or repeat core biopsy tissue sampling prior to initiation of neoadjuvant systemic chemotherapy.
* Availability of tissue blocks from initial core needle biopsy.
* Signed informed consent.
* Willing to discontinue use of all supplements containing Vitamin D for the duration of the study, and take only the Vitamin D provided by the study.

Exclusion Criteria:

* Presence of any Metastatic lesion.
* History of parathyroid disease, hypercalcemia, or kidney stones.
* History of Selective estrogen receptor modulator (SERM) or aromatase inhibitor therapy.
* Receiving metformin.
* History of renal failure requiring dialysis or kidney transplantation.
* Women who are known to be pregnant or who are nursing. (As vitamin D does not have toxicity to the fetus, a negative pregnancy test is not a requirement to participate in the study.)
* Patients planned for surgical therapy of their breast cancer or initiation of systemic chemotherapy, that would not allow for at least 7 days of vitamin D intervention
* Any condition potentially interfering with subjects ability to comply with taking study medication.
* Any medical condition that would potentially interfere with vitamin D absorption.
* Current participation in another research study that would increase risk to subject, in the opinion of the investigators.
* Patients currently taking more than 2000 IU of Vitamin D.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Telli, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Started | 25 | 16
Completed | 25 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25) | Total
Number analyzed (Participants) | 25 | 16 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 7 | 28
  >=65 years | 4 | 9 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.6) | 62.1 (7.6) | 57.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: Expression Level of Insulin-like Growth Factor-binding Protein 3 (IGFBP-3) Gene
Description: To determine whether dietary vitamin D can reverse the negative effects of obesity and insulin resistance as reflected by changes in breast cancer gene expression patterns in obese and non-obese subjects diagnosed with breast cancer. IGFBP-3 is an endocrine factors.
  Insulin-like growth factor-binding protein 3 (IGFBP-3) gene expression was assessed at baseline and after treatment in participants with body mass index (BMI) ≤ 25 and > 25. By design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day (control) and 10,000 IU/day (experimental), and is reported as the mean of the slope (a measure of magnitude of difference) between baseline and post-treatment, with standard deviation. A positive slope indicates increased expression, and a negative slope indicates decreasing values, with the larger values (positive or negative) indicating greater effect, and smaller values indicating lesser effect.
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Mean (Standard Deviation); unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | 0.02937 (0.03792) | 0.00941 (0.00680)
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | 0.0158 (0.03645) | 0.01443 (0.01828)

2. Secondary Outcome: Expression Level of Cyclin-dependent Kinase Inhibitor 1 (CDKI1; p21) Gene
Description: p21 [aka p21Cip1; p21Waf1, cyclin-dependent kinase inhibitor 1 (CDKI1) or cyclin-dependent kinase (CDK)-interacting protein 1 (CDKIP1)] gene expression was assessed at baseline and after treatment in participants with body mass index (BMI) ≤ 25 and > 25. By design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day (control) and 10,000 IU/day (experimental), and is reported as the mean of the slope (a measure of magnitude of difference) between baseline and post-treatment, with standard deviation. A positive slope indicates increased expression, and a negative slope indicates decreasing values, with the larger values (positive or negative) indicating greater effect, and smaller values indicating lesser effect.
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Mean (Standard Deviation); unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | 0.04868 (0.07735) | 0.03465 (0.03755)
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | 0.02236 (0.04859) | 0.01854 (0.01700)

3. Secondary Outcome: Expression Level of Matrix Metalloproteinase-11 (MMP-11) Gene
Description: Matrix metalloproteinase-11 (MMP-11), aka Stromelysin-3 (SL-3), gene expression was assessed at baseline and after treatment in participants with body mass index (BMI) ≤ 25 and > 25. By design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day (control) and 10,000 IU/day (experimental), and is reported as the mean of the slope (a measure of magnitude of difference) between baseline and post-treatment, with standard deviation. A positive slope indicates increased expression, and a negative slope indicates decreasing values, with the larger values (positive or negative) indicating greater effect, and smaller values indicating lesser effect.
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Mean (Standard Deviation); unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | -0.03238 (0.04776) | -0.00590 (0.02441)
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | -0.00986 (0.05814) | -0.02139 (0.01961)

4. Other Pre Specified Outcome: Expression Level of MKI67 Gene
Description: Ki 67 gene expression was assessed at baseline and after treatment in participants with body mass index (BMI) ≤ 25 and > 25. By design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day (control) and 10,000 IU/day (experimental), and is reported as the mean of the slope (a measure of magnitude of difference) between baseline and post-treatment, with standard deviation. A positive slope indicates increased expression, and a negative slope indicates decreasing values, with the larger values (positive or negative) indicating greater effect, and smaller values indicating lesser effect.
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Mean (Standard Deviation); unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | -0.00958 (0.04108) | -0.03809 (0.02416)
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | -0.01318 (0.03231) | 0.00166 (0.01412)

5. Other Pre Specified Outcome: Expression Level of ESR1 Gene
Description: ESR1 gene expression was assessed at baseline and after treatment in participants with body mass index (BMI) ≤ 25 and > 25. By design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day (control) and 10,000 IU/day (experimental), and is reported as the mean of the slope (a measure of magnitude of difference) between baseline and post-treatment, with standard deviation. A positive slope indicates increased expression, and a negative slope indicates decreasing values, with the larger values (positive or negative) indicating greater effect, and smaller values indicating lesser effect.
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Mean (Standard Deviation); unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | 0.00526 (0.14049) | -0.02739 (0.02132)
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | -0.05757 (0.0747) | 0.01225 (0.04041)

6. Other Pre Specified Outcome: Leptin to Adiponectin Ratio (Leptin:Adiponectin) in Blood
Description: Levels in blood of leptin & adiponectin were assessed at baseline & after treatment in participants with body mass index ≤25 and >25. By protocol design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day and 10,000 IU/day. For all serum protein levels, the outcome is reported as the ratio of the baseline to post-treatment values (baseline:post-treatment) of the ratio of the mean serum levels of leptin and adiponectin, (ie, lepton:adiponectin). As a ratio of the ratio of means, the outcome is reported as a number without dispersion. The outcome value expresses the treatment effect on both leptin and adiponectin collectively, with a value <1.00 meaning that the effect on leptin levels was reduced relative to the effect on adiponectin levels, and a value >1.00 that the effect on leptin levels was increased relative to the effect on adiponectin levels, with a larger difference from 1.00 indicating a greater effect (1.00 means no measure change).
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Number; unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/d: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/d | 0.87 | 1.00
  Vitamin D 10,000 IU/d: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/d | 0.95 | 1.00

7. Other Pre Specified Outcome: HOMA-IR to Adiponectin Ratio (HOMA-IR:Adiponectin) in Blood
Description: The Homeostasis Model of Assessment-Insulin Resistance (HOMA-IR) was used to assess fasting insulin & glucose levels. HOMA-IR & adiponectin were assessed at baseline & after treatment in participants with body mass index ≤25 and >25. By protocol design, the outcome is for non-obese vs obese participants stratified between 400 & 10,000 IU/day. For all serum protein levels, the outcome is reported as the ratio of the baseline to post-treatment values (baseline:post-treatment) of the ratio of the mean serum levels of leptin & adiponectin, (ie, lepton:adiponectin). As a ratio of the ratio of means, the outcome is reported as a number without dispersion. The outcome expresses the treatment effect on HOMA-IR & adiponectin collectively, with <1.00 meaning effect on HOMA-IR levels is reduced relative to the effect on adiponectin levels, & >1.00 meaning the effect is increased relative, with a greater difference meaning greater effect (1.00 represents no measure change).
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Number; unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | 0.96 | 0.52
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | 1.35 | 0.99

8. Other Pre Specified Outcome: cRP (C-reactive Protein) to Adiponectin Ratio (cRP:Adiponectin) in Blood
Description: Levels in blood of cRP (C-reactive protein) & adiponectin were assessed at baseline & after treatment in participants with body mass index (BMI) ≤25 and >25. By protocol design, the outcome was determined for non-obese vs obese participants stratified between 400 IU/day & 10,000 IU/day. For all serum protein levels, the outcome is the ratio of the baseline to post-treatment values (baseline:post-treatment) of the ratio of the mean serum levels of leptin & adiponectin, (ie, lepton:adiponectin). As a ratio of the ratio of means, the outcome is reported as a number without dispersion. The outcome value expresses the treatment effect on cRP and adiponectin collectively, with a value < 1.00 meaning effect on cRP levels was reduced relative to the effect on adiponectin levels, and a value > 1.00 meaning effect on cRP levels was increased relative to the effect on adiponectin levels, with a larger difference from 1.00 indicating a greater effect (1.00 represents no measure change).
Time Frame: up to 6 weeks
Population: Study cohorts (non-obese vs obese) are stratified by Vitamin D dose level.
Measure: Number; unit: ratio baseline:post-treatment (slope)
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
ratio baseline:post-treatment (slope)
  Vitamin D 400 IU/day: number analyzed (Participants) | 9 | 6
  Vitamin D 400 IU/day | 0.80 | 0.83
  Vitamin D 10,000 IU/day: number analyzed (Participants) | 16 | 10
  Vitamin D 10,000 IU/day | 1.33 | 1.00

9. Other Pre Specified Outcome: Pharmacokinetics of Vitamin D Metabolite Calcitriol
Description: Blood levels (pharmacokinetics) of Vitamin D were evaluated as the blood levels of Vitamin D metabolite calcitriol (also known as 1,25-dihydroxycholecalciferol or 1,25(OH)2D) in participants receiving 400 IU/day Vitamin D. The outcome is reported as the mean calcitriol level pre-treatment and post-treatment, with standard deviation.
Time Frame: up to 6 weeks
Population: All participants are included. Pharmacokinetics results are provided for non-obese vs obese participants, stratified by dose received, and presented as the pre-treatment and post-treatment pharmacokinetic values.
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: Samples for this dose & time
Groups:
- Non-obese (Body Mass Index ≤ 25): Non-obese participants receiving Vitamin D at 400 IU/day.
  Vitamin D
- Obese (Body Mass Index > 25): Obese participants receiving Vitamin D at 400 IU/day.
  Vitamin D
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
Number analyzed (Participants) | 25 | 16
Number analyzed (Samples for this dose & time) | 50 | 32
ng/mL
  Pre-treatment, 400 IU/day: number analyzed (Participants) | 9 | 3
  Pre-treatment, 400 IU/day: number analyzed (Samples for this dose & time) | 9 | 3
  Pre-treatment, 400 IU/day | 30.44 (10.89) | 34.67 (4.62)
  Pre-treatment, 10,000 IU/day: number analyzed (Participants) | 16 | 6
  Pre-treatment, 10,000 IU/day: number analyzed (Samples for this dose & time) | 16 | 6
  Pre-treatment, 10,000 IU/day | 30.75 (8.62) | 37.17 (12.51)
  Post-treatment, 400 IU/day: number analyzed (Participants) | 9 | 3
  Post-treatment, 400 IU/day: number analyzed (Samples for this dose & time) | 9 | 3
  Post-treatment, 400 IU/day | 30.89 (7.52) | 31.67 (3.06)
  Post-treatment, 10,000 IU/day: number analyzed (Participants) | 16 | 6
  Post-treatment, 10,000 IU/day: number analyzed (Samples for this dose & time) | 16 | 6
  Post-treatment, 10,000 IU/day | 53.75 (13.82) | 59.33 (27.74)

ADVERSE EVENTS:
Arm/Group | Non-obese (Body Mass Index ≤ 25) | Obese (Body Mass Index > 25)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/16
Other Adverse Events (participants affected / at risk) | 0/25 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-obese (Body Mass Index ≤ 25) (N=25) | Obese (Body Mass Index > 25) (N=16)
Primary hyperparathyroidism (HPT) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neuroendocrine cancer of the breast, metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-obese (Body Mass Index ≤ 25) (N=25) | Obese (Body Mass Index > 25) (N=16)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Plasma chromogranin A level, elevated (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes